CLINICAL TRIAL: NCT04442867
Title: A Health-social Partnership Programme for Improving Health Self-management of Community-dwelling Older Adults: a Hybrid Effectiveness-implementation Pilot Study
Brief Title: A Health-social Partnership Programme for Improving Health Self-management of Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Clinical associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEIPS
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Healthy Aging
Keywords: hybrid effectiveness-implementation design; health-social partnership; community
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects will receive nurse-led case management supported by a social service team.The nurse, functioning as a case manager, is involved in the initial assessment of the participant using the Omaha system. After the initial assessment, the NCM will equip participants with the skills required to perform self-care in health maintenance, including self-monitoring of vital signs, medication adherence, and sources of help if needed.
  Interventions: Other: Case management
- Control group (Other): Participants in the control group will receive a monthly social control call from a trained research assistant
  Interventions: Other: Social call

INTERVENTIONS:
Other: Case management — Based on the clients' problems, individualized and specific health education such as recognition of the early signs and symptoms of an exacerbation or deterioration of disease condition, the frequency, dosage, duration of each health-promoting activity that was of therapeutic value, and the techniques required to perform these activities will be provided by the Nurse Case Manager.
  Arms: Intervention group
Other: Social call — Provide social call to participants, such as ask the participants what TV program do you like most, and how are you recently.
  Arms: Control group

SUMMARY:
Health-social partnership has been governed by regulations in many developed countries for some years. For instance, the government of United Kingdom has implemented a policy specifically designed to facilitate the discharge of older adults by collaborating health and social care workers in hospitals. The United States also formulated a policy to support the development of collaborative and multi-agency care services in community setting for helping those who are vulnerable and underserved including ethnic minorities, homeless people, and those without health insurance. While these services were shown to reduce the delays in hospital discharge and improve access to services, they were found to be health-dominated and the involvement of service users in strategic design and planning was lacking. As a result, the actual process in practice was reported to be poor and a true model of health and social care partnership was not attained. Currently in Hong Kong, health-social partnership has not yet been driven and guided by policy. It is still unknown for researchers and practitioners as how to effectively build a seamless working partnership among two different disciplines and sustain in the community to support the independent living of older adults.

DETAILED DESCRIPTION:
Introduction: There is a growing body of literature supporting the involvement of a health-social approach using complex interventions in enhancing self-care management among community-dwelling older adults. However, there is a paucity of research on how this intervention strategy implements and disseminates in a real community setting. Bridging the gap between research-based evidence and primary health policy and practice is a considerable challenge to researchers, service providers and policymakers. The present pilot study aims to test the feasibility and acceptability of an evidence-based health-management intervention programme to be incorporated into the existing community services provided in the elderly centers. Results of this pilot study will provide important information if the health-social partnership program rooted in the community is acceptable and feasible and factors that may facilitate or hinder implementation when reaching the target group of older adults dwelling in the community. The preliminary outcomes of enhancing self-management and older adults in maximizing their independence in their home environment will also be examined.

Method: The present pilot study adopts an effectiveness-implementation hybrid design and intends to 1) evaluate the effectiveness of a community-based Health-Social Partnership Programme (HSPP) and 2) explore the reach, adoption, implementation, and maintenance of adopting HSPP in the community. The potential subjects will be recruited from the member list of a community centre of the Hong Kong Lutheran social services if they are (1) aged 60 or above, and (2) cognitively competent. Subjects will receive nurse-led case management supported by a social service team. Factors that hinder or facilitate the program delivery will also be examined to determine the implementation and sustained effects of the programme. The measures include the components of RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework. Data will be collected at pre-intervention (T1), post-intervention (T2), and 3 months after intervention (T3).

Discussion: There are conventional randomized controlled trials testing the effects of community-based programs but these trial designs tend to control the contextual factors rather than incorporating the program in the real environment. Positive outcomes may have been produced in these trials but it is uncertain whether the tested intervention program can be rooted in the real life context and sustain in practice. This pilot study chooses to use the hybrid model to not only test the effectiveness but also examine the measures relating to implementation.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* cognitively competent with the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) with score ≥ 22

Exclusion Criteria:

* not communicable
* not reachable by phone
* not living at home
* bedbound
* with known psychiatric problems with recent hospitalization within last 6 months
* already engaged in structured health or social programmes
* will not stay in Hong Kong for the current three months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy | baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  The change of self-efficacy in three time-points. Self-efficacy will be measured by using the Chinese version of the General Self-efficacy Scale. The scale was validated in Chinese population and had a reliability alpha coefficient of 0.89. The scale consists of ten questions, scores ranging from 10 to 40, with higher scores representing better self-efficacy.

SECONDARY OUTCOMES:
Change in quality of life | baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Quality of life will be measured by 12-item Short Form Health Survey version 2-Chinese (HK) version. The scale has been used in numerous studies with reliability confirmed when used locally. The rating of the items ranged from 0 to 100, with 50 indicating the standardized norm score.
change in health service utilisation | baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  The outcomes of health services utilisation include the total numbers of unscheduled general out-patient department, general practitioners, emergency room, and hospital admissions and the total number of health service attendance. The information will be collected by the subjective report of participants and confirmed with the medical and attendance certificates, with good reliability

CONTACTS AND LOCATIONS:
Overall Officials: Frances KY Wong, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Lutheran Social Services, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AKC, Wong FKY, Chow KKS, Kwan DKS, Lau DYS, Lau ACK. A health-social service partnership programme for improving the health self-management of community-dwelling older adults: a hybrid effectiveness-implementation pilot study protocol. Pilot Feasibility Stud. 2023 Nov 8;9(1):184. doi: 10.1186/s40814-023-01412-0. PMID 37941087
- [Derived] Wong AKC, Wong FKY, Wong MCS, Chow KKS, Kwan DKS, Lau DYS. A community-based health-social partnership program for community-dwelling older adults: a hybrid effectiveness-implementation pilot study. BMC Geriatr. 2022 Oct 7;22(1):789. doi: 10.1186/s12877-022-03463-z. PMID 36207685